CLINICAL TRIAL: NCT01003444
Title: Muscle Biopsy Study In Healthy Subjects For Malonyl Coa Biomarker Assay Development
Brief Title: Muscle Malonyl Coa Biomarker Assay Development
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B1501004
Record Dates: First submitted 2009-10-14; First posted 2009-10-28 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2009-12

CONDITIONS: Healthy Volunteers
Keywords: Muscle biopsy Malonyl CoA Biomarker assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Experimental): Muscle biopsy in healthy volunteers
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — Collection of muscle biopsies of the vastus lateralis will be performed by a consulting specialist. The first muscle biopsy (Day 1, 2 hour) will be obtained from the vastus lateralis muscle of the non-dominant leg. The second biopsy (Day 1, 4 hour) will be obtained from the same vastus lateralis muscle on the same leg approximately 10 centimeters from the first muscle biopsy site.

SUMMARY:
Biopsies of the outer thigh muscle and serum samples will be collected from untreated healthy subjects. These biological samples will be provided to the Diabetes Research Unit Translational Biomarker Laboratory for use in developing and validating human muscle malonyl CoA and serum malonate biomarker assays.

DETAILED DESCRIPTION:
This non-drug method study was terminated on November 19, 2009. The decision to terminate was based on safety concerns (biopsy-related pain) observed in the first set of subjects. Four subjects were give a sample and did not tolerate it well. No data was collected to report.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests). Female subjects will be of non-childbearing potential.
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, allergic, (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing), muscle disease, diabetes, or severe uncontrolled hypertension.
* Any significant bleeding diathesis which could preclude recovery from the biopsy procedure. ASA, ibuprofen, and any other oral anti platelet agent should be discontinued at least 7 days prior to procedure.
* Prothrombin time (PT)/INR and/or activated partial thromboplastin time (aPTT) above the respective local laboratory normal ranges.
* Abnormal CK as per CRU laboratory ranges.
* Subjects with either a medical history of or physical evidence of keloid scar formation upon physical examination.
* 12 lead ECG demonstrating a clinically significant abnormality.
* Females of child bearing potential, pregnant or nursing females or females less than 6 months postpartum from the scheduled date of collection.
* Known hypersensitivity to lidocaine or any component of the study procedure.
* Participation in non-routine rigorous exercise (eg, road races, heavy lifting, etc.) within one week prior to the muscle biopsy procedures.
* Professional athletes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Vastus lateralis skeletal muscle samples (>=100 mg but not to exceed 300 mg) will be collected from 12 healthy subjects for provision to the Diabetes Research Unit Translational Biomarker Laboratory. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1501004&StudyName=Muscle%20Malonyl%20Coa%20Biomarker%20Assay%20Development